CLINICAL TRIAL: NCT01768585
Title: A Randomised, Placebo Controlled, Double Blind, Cross-over, Single Center Clinical Study to Investigate the Effect of Heart Rate Reduction With Ivabradine on Vascular Elastic Properties and Endothelial Function in Patients With Stable Coronary Heart Disease
Brief Title: Study to Investigate the Effect of Heart Rate Reduction With Ivabradine on Vascular Elastic Properties and Endothelial Function in Patients With Stable Coronary Heart Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Saarland (Other)
Collaborators: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HomRate04_2012
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease; Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivabradine (Active Comparator): Drug: Ivabradine bid administration of 7.5mg ivabradine Other Name: Procoralan, I(f)-inhibitor
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator): Drug: Placebo bid placebo Other Name: Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — Please see description of Intervention Arm
  Other Names: Procoralan
  Arms: Ivabradine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study investigates whether chronic heart rate reduction with ivabradine (Procoralan®, Servier, France) affects aortic compliance and endothelial function in patients with chronic stable coronary artery disease.

DETAILED DESCRIPTION:
Experimental and clinical data suggest that sustained elevation of heart rate contributes to the pathogenesis of vascular disease (1, 2). In animal studies accelerated heart rate is associated with signalling events leading to vascular oxidative stress, endothelial dysfunction and acceleration of atherogenesis (3). The underlying mechanisms are only partially understood and appear to correlate with mechanic properties such as reduction of vascular compliance. Heart rate reduction by I(f)-channel inhibition with ivabradine (Procoralan®, Servier, France) attenuates oxidative stress, improves endothelial function and reduces the formation of atherosclerotic plaques in mice models of lipid-induced atherosclerosis (1, 4).

Aortic stiffness is a consequence of arterial aging and vascular risk factors and determinates cardiovascular mortality (5). Heart rate depending repetitive pulsations appear to induce fatigue and fracture of elastin lamellae of central arteries. As a result the vessel stiffens and pulse wave reflections return earlier to the heart. In consequence aortic pressure rises and pulsations of flow extend further into smaller vessels of organs (notably the brain and kidney). Stiffening leads to increased left ventricular (LV) load with hypertrophy, decreased capacity for myocardial perfusion, and increased hemodynamic stresses on small arterial vessels.

Several experimental investigations revealed an interaction between heart rate and vascular compliance demonstrating a positive association between increased heart rate and arterial stiffness (6). Recent experimental data suggest that heart rate reduction by ivabradine (Procoralan®, Servier, France) significantly improves aortic distensibility in cholesterol fed ApoE -/- mice measured by MRI technique (7). While a benefit of pharmacological heart rate reduction on vascular outcomes was observed in animal studies, prospective clinical data are limited and evidence determining whether chronic modulation of heart rate can improve vascular function and compliance in patients with chronic stable coronary artery disease is needed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Resting heart rate ≥ 70 bpm
* Sinus rhythm
* Chronic stable coronary artery disease (CAD)
* Coronary artery disease proven by coronary angiography
* Written informed consent to participate in the study

Exclusion Criteria:

* Acute coronary syndrome
* CAD treated best by surgical coronary bypass
* Stroke/TIA
* Resting heart rate < 70 bpm
* Indwelling pacemaker or AICD
* Severe valvular heart disease
* Any other rhythm than sinus
* Sick-Sinus-Syndrome, SA nodal block, >2nd degree atrio-ventricular block
* Untreated arterial hypertension
* Arterial hypotension (<90/50mmHg)
* Severe hepatic failure
* Heart failure (NYHA class III - IV)
* Patient already treated with study drug
* Symptomatic PAD
* Known diabetes mellitus
* Pre-menopausal women
* Hypersensitivity against ivabradine or adjuvants
* Coexisting drug treatment with Cytochrom P450 3A4-inhibitors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Aortic distensibility (MRI), pulse wave velocity (SphygmoCor®), flow-mediated dilatation (A. brachialis) | Decembre 2014

SECONDARY OUTCOMES:
Biomarkers (inflammation, oxidative stress) | Decembre 2014

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Laufs, Principal Investigator — Saarland University Hospital
Locations (1):
- University Hospital, Saarland, Homburg, Saarland, Germany

REFERENCES:
- [Background] Custodis F, Baumhakel M, Schlimmer N, List F, Gensch C, Bohm M, Laufs U. Heart rate reduction by ivabradine reduces oxidative stress, improves endothelial function, and prevents atherosclerosis in apolipoprotein E-deficient mice. Circulation. 2008 May 6;117(18):2377-87. doi: 10.1161/CIRCULATIONAHA.107.746537. Epub 2008 Apr 28. PMID 18443241
- [Background] Beere PA, Glagov S, Zarins CK. Retarding effect of lowered heart rate on coronary atherosclerosis. Science. 1984 Oct 12;226(4671):180-2. doi: 10.1126/science.6484569.
- [Background] Custodis F, Schirmer SH, Baumhakel M, Heusch G, Bohm M, Laufs U. Vascular pathophysiology in response to increased heart rate. J Am Coll Cardiol. 2010 Dec 7;56(24):1973-83. doi: 10.1016/j.jacc.2010.09.014. PMID 21126638
- [Background] Noels H, Weber C. Fractalkine as an important target of aspirin in the prevention of atherogenesis : Editorial to: "Aspirin inhibits fractalkine expression in atherosclerotic plaques and reduces atherosclerosis in ApoE gene knockout mice" by H. Liu et al. Cardiovasc Drugs Ther. 2010 Feb;24(1):1-3. doi: 10.1007/s10557-009-6213-4. No abstract available. PMID 20033269
- [Background] Cavalcante JL, Lima JA, Redheuil A, Al-Mallah MH. Aortic stiffness: current understanding and future directions. J Am Coll Cardiol. 2011 Apr 5;57(14):1511-22. doi: 10.1016/j.jacc.2010.12.017. PMID 21453829
- [Background] Mangoni AA, Mircoli L, Giannattasio C, Ferrari AU, Mancia G. Heart rate-dependence of arterial distensibility in vivo. J Hypertens. 1996 Jul;14(7):897-901. doi: 10.1097/00004872-199607000-00013. PMID 8818929
- [Background] Custodis F, Fries P, Muller A, Stamm C, Grube M, Kroemer HK, Bohm M, Laufs U. Heart rate reduction by ivabradine improves aortic compliance in apolipoprotein E-deficient mice. J Vasc Res. 2012;49(5):432-40. doi: 10.1159/000339547. Epub 2012 Jul 3. PMID 22759927